CLINICAL TRIAL: NCT01904110
Title: For 12months, the Multi Center, Randomized, Open-label Comparative Clinical Study to Evaluate the Efficacy and the Safety of Monthly(RisenexM Group) Versus Weekly Oral Risedronate(Risenexsplus Group) With Vitamin D in Compliance, Improvement of Vitamin D and BMD in Korean Postmenopausal Osteoporotic Women(Phase IV)
Brief Title: To Evaluate the Efficacy and the Safety of Monthly Versus Weekly Oral Risedronate With Vitamin D in Compliance, Improvement of Vitamin D and BMD in Korean Postmenopausal Osteoporotic Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL_RSNM_401
Record Dates: First submitted 2013-07-16; First posted 2013-07-22 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Osteoporosis
Keywords: Risedronate,cholecalciferol,BMD,montly,weekly,compliance
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risenex M (Experimental): Patients who were treated with Resenex M (Risendronate/Cholecalciferol combination in one tablet) once a month for 12months
  Interventions: Drug: Risedronate/Cholecalciferol combination(montly)
- Risenex Plus (Active Comparator): Patients who were treated with Risenex plus (Risendronate/Cholecalciferol combination in one tablet) once a week for 12months
  Interventions: Drug: Risedronate/Cholecalciferol combination(montly); Drug: Risedronate/Cholecalciferol combination(weekly)

INTERVENTIONS:
Drug: Risedronate/Cholecalciferol combination(montly) — once a month
  Other Names: Risenex M
Drug: Risedronate/Cholecalciferol combination(weekly) — once a week
  Other Names: Risenex Plus
  Arms: Risenex Plus

SUMMARY:
The purpose of this study is to evaluate the Efficacy and the Safety of Monthly(RisenexM group) versus Weekly Oral risedronate(Risenexsplus group) in Korean postmenopausal osteoporotic women(Phase IV)

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Efficacy and the Safety of Monthly(RisenexM group) versus Weekly Oral risedronate(Risenexsplus group) with Vitamin D in compliance, improvement of vitaminD and BMD in Korean postmenopausal osteoporotic women(Phase IV)

ELIGIBILITY:
Inclusion Criteria:

1. Female osteoporosis patients over 19years of age(with menopause).

   Definition of osteporosis
   * They had a BMD T-score -2.5 or less at mean Lumbar spine(L1~L4), Femoral neck or total. Or evidence of at least one vertebral fracture.

   Definition of menopause(can be one of three condition)
   * For 12months spontaneous amenorrhea
   * For 6months spontaneous amenorrhea with serum FSH(Follicle stimulating hormone) is 40 mlIU/mL and over
   * 6weeks after bilateral ovariectomy whether hysterectomy of not
2. Patients who can be treated with oral bisphosphonate drugs
3. Patients who have adequate to be measured DXA(Dual energy x-ray absorptiometry)
4. Patients who made a voluntary agreement after explanation of this study
5. Patients who participated in clinical trial(HL_RSNP_401) must have taken the Risenexplus and finish the study for 12 months.

Exclusion Criteria:

1. Patients with esophagus disorder.
2. Patients administered with osteoprosis therapy(except calcium,Vit.D medication) within previous 3 months
3. Patients with serum calcium concentrations 8.0mg/dL under.
4. Patients with severe nephropathy(serum creatinine> doulble of normal level
5. Patients with unable to sit upright or stand 30minutes.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05-29 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
The propotion of patients with 25(Oh)D level <20mg/ml of 12 months | 1 year

SECONDARY OUTCOMES:
The change of Bone Mineral Density(BMD) value | 1year
  The change of Bone Mineral Density(BMD) value[Time frame: 1 year] The change of PTH(Parathyroid hormone value) [Time frame:6months,1 year] The change of Compliance - overall groups of Risenex plus vs Risenex M(2groups)
The change of PTH(Parathyroid hormone value) | 6months,1 year
  The change of Bone Mineral Density(BMD) value[Time frame: 1 year] The change of PTH(Parathyroid hormone value) [Time frame:6months,1 year] The change of Compliance - overall groups of Risenex plus vs Risenex M(2groups)
The change of Compliance - overall groups of Risenex plus vs Risenex M | 1year
  The change of Bone Mineral Density(BMD) value[Time frame: 1 year] The change of PTH(Parathyroid hormone value) [Time frame:6months,1 year] The change of Compliance - overall groups of Risenex plus vs Risenex M(2groups
The change of 25(Oh)D level in patients. | 6months,1year

CONTACTS AND LOCATIONS:
Overall Officials: Youngki Min, MD, Principal Investigator — Samsung Medical Center Seoul
Locations (1):
- Samsung Medical Center, Seoul, South Korea